CLINICAL TRIAL: NCT04269616
Title: The Effect of Order of Presenting Survival and Disability Information for Periviable Births on Participant Treatment Choice
Brief Title: Order Effects of Prematurity Outcome Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 2019-121
Record Dates: First submitted 2020-02-07; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Premature Birth
Keywords: Decision making; Neonatal resuscitation; Order effect; Prenatal counseling
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: 2x2 between subjects
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Numerical survival, followed by disability information (Experimental): Participants in this arm were presented with a pictograph displaying numerical survival information, followed by a pictograph displaying disability information.
  Interventions: Behavioral: Order of pictographs provided to participants; Behavioral: Level of description in survival pictograph
- Survival with description, followed by disability information (Experimental): Participants in this arm were presented with a pictograph displaying survival information including the average course of stay in the NICU, followed by a pictograph displaying disability information.
  Interventions: Behavioral: Order of pictographs provided to participants; Behavioral: Level of description in survival pictograph
- Disability information, followed by numerical survival (Experimental): Participants in this arm were presented with a pictograph displaying disability information, followed by a pictograph displaying numerical survival.
  Interventions: Behavioral: Order of pictographs provided to participants; Behavioral: Level of description in survival pictograph
- Disability information, followed by survival with description (Experimental): Participants in this arm were presented with a pictograph displaying disability information, followed by a pictograph displaying survival information including the average course of stay in the NICU.
  Interventions: Behavioral: Order of pictographs provided to participants; Behavioral: Level of description in survival pictograph

INTERVENTIONS:
Behavioral: Order of pictographs provided to participants — The pictographs presented to participants about survival and disability were varied in the order in which they were presented (i.e. survival or disability information first).
Behavioral: Level of description in survival pictograph — The pictographs presented to participants about survival and disability were varied in the level of description provided in the survival pictograph (i.e. only numerical data, or also a description of course of NICU stay).

SUMMARY:
Women recruited from the internet were put in a hypothetical situation of being in labor at 22 weeks of pregnancy, and presented with information in the form of pictographs about survival and disability of babies born at this gestational age.

Participants were randomized to receive these pictographs in a different order (survival or disability first) and to receive descriptiveness level of survival (just numerical information, or also description of course of NICU stay).

Participants were then asked to choose between comfort care and intensive care in this situation. Participants' religiosity, value of the sanctity of life, and health literacy were also assessed.

DETAILED DESCRIPTION:
The National Institute of Child Health and Human Development (NICHD) Workshop on Periviable Birth recommended that information on the chance of survival and risk of disability should be provided separately. The order in which information is presented can affect memory, persuasiveness, and treatment choice, but the effect of order of information presentation in the context of neonatal resuscitation has received little attention. Additionally, the effect of including a description of the long and intense time in the neonatal intensive care unit (NICU) on parental treatment decision making is also unexplored. Current evidence suggests that pictographs best convey numerical information to parents.

Three pictographs were developed based on NICHD data for 22 weeks gestational age (GA) babies who received intensive care. One pictograph displayed information on the rates of disability in the babies who survive. Two pictographs displayed information about how many babies born at 22 weeks survive, with one of these pictographs including a description of the average course of NICU stay.

An internet survey was sent to a U.S. representative sample of women of child-bearing age. A vignette including background on prematurity and the treatment options of intensive care or comfort care for a baby born at 22 weeks GA was presented. Participants viewed the pictographs, evenly randomized to one of four experimental conditions (order of information presentation x level of description of NICU course). Participants were then asked to choose intensive care or comfort care. Participant religiosity, values (quality vs. sanctity of life), autonomy preferences in medical decision making, previous NICU exposure, numeracy, and health literacy were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing age (defined as 18-50) living in the U.S.

Exclusion Criteria:

* Minors, those unable to read English, and those who only could complete the survey on their phone. (For formatting purposes, a tablet or computer was necessary.)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The survey was distributed only to women.
Enrollment: 839 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
Hypothetical treatment choice | Assessed immediately post-intervention.
  Participant's hypothetical treatment choice of either comfort care or intensive care. Participants were told: "Your doctor asks you what treatment option you want to choose," and given the options of "I would want the doctors to provide the baby intensive care / comfort care." This dichotomous variable is assessed for the frequency of each option chosen.

SECONDARY OUTCOMES:
Religiosity | Assessed post-intervention, immediately after treatment choice.
  Participants' religiosity was assessed using the Duke University Religion Index (5-item). Potential scores range from 5-27, with 27 being the most religious.
Preference for medical autonomy | Assessed post-intervention, immediately after treatment choice.
  Participants were asked on a 4-point scale their medical autonomy preferences, in the form of: "In making medical decisions: 1) I always prefer to have the doctor make decisions for me, 2) I would prefer to have the doctor make medical decisions for me most of the time, 3) I would prefer to make my own medical decisions most of the time, or 4) I always prefer to make my own decisions." Score ranging from 1-4, with 4 being the maximum preference for medical autonomy.
Values: quality or sanctity of life | Assessed post-intervention, immediately after treatment choice.
  Participants answered the following: "In making end-of-life decisions: 1) Quality of life is much more important than preserving life, 2) Quality of life is somewhat more important than preserving life, 3) Preserving life is somewhat more important than quality of life, or 4) Preserving life is much more important than quality of life." In the range of 1-4, a score of 4 indicated the greatest participant value of sanctity of life.
Numeracy | Assessed post-intervention, immediately after treatment choice.
  Participants' numeracy levels were assessed by using an adapted item from the Subjective Numeracy Scale: "How good are you at figuring out how much a $20 shirt will cost if it is 25% off? Extremely / Quite a bit / Somewhat / A little bit / Not at all." Participants who answered somewhat, a little bit, or not at all were considered to have low numeracy.
Health literacy | Assessed post-intervention, immediately after treatment choice.
  Participants' health literacy was assessed using the single-item Brief Health Literacy screening, which asks, "How confident are you filling out medical forms by yourself? Extremely / Quite a bit / Somewhat / A little bit / Not at all." Participants who answered somewhat, a little bit, or not at all were considered to have low health literacy.
Previous NICU exposure | Assessed post-intervention, immediately after treatment choice.
  Participants were also asked if they have previously had a child in the NICU, with yes/no answer options.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States